CLINICAL TRIAL: NCT06668740
Title: The Influence of Using Virtual Reality Glasses on the Quality of Life of the Elderly
Brief Title: Evaluation of a Program to Improve the Life Quality of Elderly
Acronym: VR_LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Dèlia Borda Fortuny, Nurse, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23/155-P
Record Dates: First submitted 2024-09-18; First posted 2024-10-31 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Elderly
Keywords: VirtualReality; Quality of Life; Elderly
MeSH Terms: interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): A pretest was conducted with a group of elderly residents from three different nursing homes. Following this, participants watched 360-degree VR videos featuring nature walks, trips, and similar experiences for 10 minutes, once a week, over a period of four weeks. After completing the VR sessions, a posttest was administered. The results will be used to assess the participants' Quality of Life and their Satisfaction with the intervention.
  Interventions: Behavioral: The use of Virtual Reality Glasses in Elderly

INTERVENTIONS:
Behavioral: The use of Virtual Reality Glasses in Elderly — The group first completed a pretest, after which they watched 360-degree VR videos, such as nature walks and trips, for 10 minutes once a week over four weeks. Following this, a posttest was conducted. The outcomes will be used to measure changes in Quality of Life.

SUMMARY:
Older people belong to an age group that has been increasing in recent decades, leading to a progressive ageing of the population. With the aim of reducing the generational digital divide, the use of technology in retirement homes was proposed. To this end, virtual reality glasses were used to allow the visualization of an external virtual world and, subsequently, it was evaluated whether their application improved the quality of life of the elderly by reducing the difficulties they have in participating in recreational activities outside these centers. A prospective quasi-experimental longitudinal study was carried out in the centers belonging to the basic health area of Valls, with a study period from May 2023 to March 2024. Quality of life was measured using the ad hoc "Escala de Calidad de Vida Rivas-Bordas".

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older.
* Resident of a geriatric home in the Valls area.
* Individuals with slight, moderate, fair, or total impairment of social resources, as assessed by the Duke University Center (1978) Social Resources Scale (OARS).

Exclusion Criteria:

* Individuals with a history of frequent migraines or motion sickness.
* Individuals with moderate or severe cognitive impairment (≥ 5 errors on the Abbreviated Pfeiffer test).
* Inability to communicate in Spanish and/or Catalan.
* Individuals with advanced visual and/or hearing impairments.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Level of Quality of Life | pre-intervention and immediately after post-intervention
  The Quality of Life was evaluated using the ad hoc "Rivas-Borda Quality of Life Scale." Developed by the principal investigators, it consists of 26 items. The scale measures participants' Quality of Life across four areas (emotional, cognitive, socio-economic, and physical) using a 4-point Likert scale (1 = Never or almost never, 4 = Always or almost always). The lowest possible score on the scale is 23, and the highest is 104. A score between 104 and 81 indicates an adequate Quality of Life, between 80 and 54 points suggests a risk of Quality of Life deterioration, and between 53 and 23 indicates an altered Quality of Life.
  At the end of the scale, there are 3 additional questions assessing satisfaction with the activity, also rated on a 4-point Likert scale (1 = Not at all, 4 = Very much).

SECONDARY OUTCOMES:
Gender | pre-intervention
  Female, Male or Non-binary
Marital Statuts | pre-intervention
  Single, widowed, married or in a partner living in the residence or married or in a partner who does not live in the residence.

CONTACTS AND LOCATIONS:
Locations (1):
- Delia Borda Fortuny, Bellcaire d'Urgell, Lleida, Spain